CLINICAL TRIAL: NCT03508284
Title: Factors Associated With Dual-Task Performance in Patients With Multiple Sclerosis
Brief Title: Dual-Task Performance in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Other Study IDs: 230
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Dual-task; Balance; Mobility; Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: MS patients (EDSS: 0-5,5)
- Healthy group: Healthy individuals without chronic disease

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory disease affecting the central nervous system. It is reported that 85% of patients with multiple sclerosis have gait disturbance, 88% balance, and 35-90% fatigue (1, 2, 3). In addition, 65% of patients are reported that their cognitive functions have regressed (4).

It is important to increase the independence of the MS patients in activities of daily living (ADL). Almost all of ADL requires many activities at the same time. For example, toothbrushing involves both the standing balance and the motor activity of the upper limb at the same time. It also requires cognitive tasks such as attention and focusing. Many activities that seem to be the only task are actually multitasking (5).

The aim of this study is to investigate the effects of motor and cognitive additional task on balance, mobility and upper limb performances in MS patients and to determine the factors associated with dual-task performance.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The balance, mobility, upper extremity performance, cognitive function, fatigue, physical activity level, mood, sleep quality, quality of life will be evaluated once.

We will use descriptive statistics and t-tests to compare demographic characteristics between groups and for the categorical variables chi-square. Effect of the group (MS patients or healthy controls), condition (Single task and dual-task conditions), and group × condition interaction will be compared using two-way repeated measures ANOVA. We will examine the correlations between fatigue severity, physical activity level, mood, sleep quality, quality of life using Pearson bivariate correlations. The significance level is set at p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who 18-65 years of age
* MS patients who are ambulatory (Expanded Disability Status Scale score ≤ 5,5 ) in a stable phase of the disease, without relapses in the last 3 month.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients who apply to the Neurological Rehabilitation Unit of Gazi University Faculty of Health Sciences will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | ten minutes
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
  Cognitive additional task (arithmetic): Individuals will be asked to perform tasks by counting backward from 3 to 3 from 100.
  Cognitive additional task (verbal): Individuals will be asked to fulfill their duties by producing a vegetable-fruit name.
Modified Sensory Organization Test | Fifteen minutes
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.
  * Cognitive additional task (arithmetic)
  * Cognitive additional task (verbal)
upper extremity function | ten minutes
  9-Hole Peg Test
  * Cognitive additional task (arithmetic)
  * Cognitive additional task (verbal)

SECONDARY OUTCOMES:
Sleep Quality: PSQI | 5-10 minutes
  The Pittsburgh Sleep Quality Index (PSQI) assess sleep quality. It is completed in 5-10 minutes. It consists of seven subscales: subjective sleep efficiency, sleep latency, sleep duration, sleep quality, sleep disturbance, sleep medication use, and daytime dysfunction due to sleepiness. Subscales yield a score from 0 to 3 and PSQI total score of >5 is indicative of poor sleep.
Fatigue Severity | Five minutes
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.
Balance Confidence | five minutes
  Activities-specific Balance Confidence (ABC) is a scale in which the patient rates his perceived level of confidence while performing 16 daily living activities.
Mood | one minute
  Beck's Depression Inventory
Visual attention and task switching | Five minutes
  Trail Making Test
selective attention | Five minutes
  stroop test
cognitive function | thirty minutes
  The Brief Repeatable Battery of Neuropsychological Tests

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebert JR, Corboy JR. The association between multiple sclerosis-related fatigue and balance as a function of central sensory integration. Gait Posture. 2013 May;38(1):37-42. doi: 10.1016/j.gaitpost.2012.10.015. Epub 2012 Nov 28. PMID 23200463
- [Background] Mostert S, Kesselring J. Effects of a short-term exercise training program on aerobic fitness, fatigue, health perception and activity level of subjects with multiple sclerosis. Mult Scler. 2002 Apr;8(2):161-8. doi: 10.1191/1352458502ms779oa. PMID 11990874
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Background] Kalron A, Dvir Z, Achiron A. Walking while talking--difficulties incurred during the initial stages of multiple sclerosis disease process. Gait Posture. 2010 Jul;32(3):332-5. doi: 10.1016/j.gaitpost.2010.06.002. Epub 2010 Jul 1. PMID 20594850
- [Background] Yelnik A, Bonan I. Clinical tools for assessing balance disorders. Neurophysiol Clin. 2008 Dec;38(6):439-45. doi: 10.1016/j.neucli.2008.09.008. Epub 2008 Oct 18. PMID 19026963
- [Background] Hofheinz M, Mibs M. The Prognostic Validity of the Timed Up and Go Test With a Dual Task for Predicting the Risk of Falls in the Elderly. Gerontol Geriatr Med. 2016 Mar 16;2:2333721416637798. doi: 10.1177/2333721416637798. eCollection 2016 Jan-Dec. PMID 28138492
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Kaya Y, Aki OE, Can UA, Derle E, Kibaroglu S, Barak A. Validation of Montreal Cognitive Assessment and Discriminant Power of Montreal Cognitive Assessment Subtests in Patients With Mild Cognitive Impairment and Alzheimer Dementia in Turkish Population. J Geriatr Psychiatry Neurol. 2014 Jun;27(2):103-9. doi: 10.1177/0891988714522701. Epub 2014 Feb 26. PMID 24578463
- [Background] Boringa JB, Lazeron RH, Reuling IE, Ader HJ, Pfennings L, Lindeboom J, de Sonneville LM, Kalkers NF, Polman CH. The brief repeatable battery of neuropsychological tests: normative values allow application in multiple sclerosis clinical practice. Mult Scler. 2001 Aug;7(4):263-7. doi: 10.1177/135245850100700409. PMID 11548987
- [Background] Benedict RH, Munschauer F, Linn R, Miller C, Murphy E, Foley F, Jacobs L. Screening for multiple sclerosis cognitive impairment using a self-administered 15-item questionnaire. Mult Scler. 2003 Feb;9(1):95-101. doi: 10.1191/1352458503ms861oa. PMID 12617275
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Idiman E, Uzunel F, Ozakbas S, Yozbatiran N, Oguz M, Callioglu B, Gokce N, Bahar Z. Cross-cultural adaptation and validation of multiple sclerosis quality of life questionnaire (MSQOL-54) in a Turkish multiple sclerosis sample. J Neurol Sci. 2006 Jan 15;240(1-2):77-80. doi: 10.1016/j.jns.2005.09.009. Epub 2005 Nov 8. PMID 16277993